CLINICAL TRIAL: NCT01601665
Title: Post Approval Study of the AcrySof® IQ Toric High Cylinder Power IOL Models SN6AT6-SN6AT9
Brief Title: Post Approval Study of the AcrySof® IQ Toric Intraocular Lens (IOL) Models SN6AT6-SN6AT9
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: C-11-020
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Cataracts; Astigmatism
Keywords: Intraocular lens; Cataracts; Astigmatism; Toric
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Toric High Cylinder Power IOL: Toric high cylinder power intraocular lens implanted during cataract surgery in the first operative eye, with the second operative eye implanted within 30 days of the first implantation.
  Interventions: Device: SN6AT6 Intraocular Lens; Device: SN6AT7 Intraocular Lens; Device: SN6AT8 Intraocular Lens; Device: SN6AT9 Intraocular Lens
- Monofocal IOL: Monofocal intraocular lens implanted during cataract surgery in the first operative eye, with the second operative eye implanted within 30 days of the first implantation.
  Interventions: Device: SN60WF Intraocular Lens

INTERVENTIONS:
Device: SN6AT6 Intraocular Lens — Acrylic intraocular lens with cylinder power at the IOL plane of 3.75 diopters. Intraocular lenses are implanted during cataract surgery as a replacement for the natural crystalline lens and are intended for long term use over the lifetime of the cataract subject.
  Other Names: AcrySof® IQ Toric Model SN6AT6
  Groups: Toric High Cylinder Power IOL
Device: SN6AT7 Intraocular Lens — Acrylic intraocular lens with cylinder power at the IOL plane of 4.50 diopters. Intraocular lenses are implanted during cataract surgery as a replacement for the natural crystalline lens and are intended for long term use over the lifetime of the cataract subject.
  Other Names: AcrySof® IQ Toric Model SN6AT7
  Groups: Toric High Cylinder Power IOL
Device: SN6AT8 Intraocular Lens — Acrylic intraocular lens with cylinder power at the IOL plane of 5.25 diopters. Intraocular lenses are implanted during cataract surgery as a replacement for the natural crystalline lens and are intended for long term use over the lifetime of the cataract subject.
  Other Names: AcrySof® IQ Toric Model SN6AT8
  Groups: Toric High Cylinder Power IOL
Device: SN6AT9 Intraocular Lens — Acrylic intraocular lens with cylinder power at the IOL plane of 6.00 diopters. Intraocular lenses are implanted during cataract surgery as a replacement for the natural crystalline lens and are intended for long term use over the lifetime of the cataract subject.
  Other Names: AcrySof® IQ Toric Model SN6AT9
  Groups: Toric High Cylinder Power IOL
Device: SN60WF Intraocular Lens — Acrylic aspheric monofocal intraocular lens. Intraocular lenses are implanted during cataract surgery as a replacement for the natural crystalline lens and are intended for long term use over the lifetime of the cataract subject.
  Other Names: AcrySof® IQ Aspheric NATURAL Model SN60WF
  Groups: Monofocal IOL

SUMMARY:
The purpose of this study is to evaluate the use of toric high cylinder power intraocular lenses in a larger population in clinical practice and assure the continued safety of these approved devices.

DETAILED DESCRIPTION:
In this prospective, non-randomized, unmasked study, subjects with pre-existing corneal astigmatism ≥2.57 diopters will choose to be implanted with either the AcrySof® IQ Toric High Cylinder Power IOL or the AcrySof® IQ Aspheric NATURAL monofocal IOL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bilateral cataracts and in the targeted astigmatism range.
* Planned cataract removal by phacoemulsification.
* Pupil size greater than or equal to 6 mm after dilation.
* Able to undergo second eye surgery within 30 days of first eye surgery.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Irregular corneal astigmatism.
* Any inflammation or swelling of the cornea.
* Any corneal abnormality other than regular corneal astigmatism.
* Previous corneal refractive surgery.
* Amblyopia.
* Diabetic retinopathy.
* Uncontrolled glaucoma.
* Currently participating in another investigational drug or device study that may confound the results of this investigation.
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be selected from up to 80 clinical investigative sites.
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Rate of Severe Visual Distortions | 6 months
  As assessed by a Patient Reported Outcomes (PRO) questionnaire. Subjects will be categorized as experiencing a severe visual distortion if they indicate "severe" as a response to any of the three visual distortion-related questions on the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Calderon, CM, Surgical, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

REFERENCES:
- [Derived] Holladay JT, Wilcox RR, Koch DD, Wang L. Astigmatism analysis and reporting of surgically induced astigmatism and prediction error. J Cataract Refract Surg. 2022 Jul 1;48(7):799-812. doi: 10.1097/j.jcrs.0000000000000871. PMID 35749069